CLINICAL TRIAL: NCT02006199
Title: Effect of Mindfulness Based Treatment for Obsessive-compulsive Disorder
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Withdrawal of the administrative reason
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 1306-076-498
Record Dates: First submitted 2013-12-04; First posted 2013-12-10 (Estimated); Last update posted 2016-10-14 (Estimated); Status verified 2013-12

CONDITIONS: Obsessive-compulsive Disorder
Keywords: obsessive-compulsive disorder; mindfulness; meditation
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Mindfulness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- relaxation with psychoeducation (Experimental): after 8 weeks of relaxation with psychoeducation. subject take part in 8 weeks of the mindfulness meditation program
  Interventions: Behavioral: mindfulness meditation
- meditation (Experimental): 8 weeks of mindfulness meditation
  Interventions: Behavioral: mindfulness meditation

INTERVENTIONS:
Behavioral: mindfulness meditation — 8 weeks of mindfulness meditation specified for OCD patient

SUMMARY:
Hypothesis of this study is that mindfulness meditation would decrease the severity of obsessive-compulsive symptoms.

DETAILED DESCRIPTION:
Before and after 8 weeks of mindfulness program, We will measure Y-BOCS scores in OCD patients. As a control program, relaxation and psychoeducation will provided to OCD patients.

ELIGIBILITY:
Inclusion Criteria:

* obsessive-compulsive disorder
* age 17-55

Exclusion Criteria:

* currently undergoing Cognitive Behavioral Therapy, psychotherapy
* other medical disease

Ages: 17 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2013-10; Primary Completion 2014-07 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
Yale-Brown Obsessive compulsive scores | 8 weeks

SECONDARY OUTCOMES:
Neurocognitive profile (emotion-memory task) | 8 weeks

OTHER OUTCOMES:
HAM-D | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jun Soo Kwon, MD phD, Principal Investigator — Seoul National University College of Medicine
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No